CLINICAL TRIAL: NCT04852458
Title: Glucocorticoids After Traumatic Birth and the Associated Risk of Developing Posttraumatic Stress Disorder (PTSD): an Open Label Pilot Trial
Brief Title: Glucocorticoid Administration After Traumatic Birth
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Joanna Kountanis, Assistant Professor of Anesthesiology and Assistant Professor of Obstetrics and Gynecology, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00174658
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Traumatic Birth
Keywords: Posttraumatic stress disorder
MeSH Terms: conditions — Birth Injuries; Stress Disorders, Post-Traumatic | interventions — Hydrocortisone; hydrocortisone hemisuccinate

STUDY DESIGN:
Intervention Model Description: There will be an observation cohort, from which individuals who can be approached within the critical time thresholds and who meet inclusion criteria will be invited to join an open label treatment arm.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous hydrocortisone (Experimental)
  Interventions: Drug: Intravenous (IV) hydrocortisone
- Observational (No Intervention): Participants will complete assessments/surveys only.

INTERVENTIONS:
Drug: Intravenous (IV) hydrocortisone — Participants (20) will be given IV hydrocortisone within 6-12 hours of the traumatic event.
  90 - 150 mg. of intravenous hydrocortisone dosing regimen based on participant weight: 90mg will be administrated to participants weighing 45-59kg. 100mg will be administrated to participants weighing 60-69kg. 120mg will be administrated to participants weighing 70-89kg. 140mg will be administrated to participants weighing 90-99kg. 150mg will be administrated to participants weighing 100-120kg.
  Other Names: Solu-Cortef®
  Arms: Intravenous hydrocortisone

SUMMARY:
This study has two components, an observational and a trial component. The observational part is being done to screen for postpartum posttraumatic stress disorder by collecting mental health assessments in women who are immediately postpartum for up to 6 weeks.

Additionally, the project has a small number of subjects that will participate in a clinical trial in which they would self-select to receive one dose of hydrocortisone intravenously while they are in the hospital. This pilot of up to 20 participants in the trial arm is designed to create a first indication of whether this could become an effective early intervention to prevent PTSD if given while trauma memories are first being formed.

This registration will list the observational part (number of participants =100) as well as the clinical trial (number of participants =20).

ELIGIBILITY:
Inclusion Criteria (for observation and hydrocortisone treatment groups):

* Screening positive for PTSD Diagnostic and Statistical Manual of Mental Disorders-5 Criteria A (felt a threat to life or injury to self or neonate)
* Postpartum hemorrhage or emergency cesarean delivery
* Owner of a smart phone or email account

Exclusion Criteria (for observation and hydrocortisone treatment groups):

* Active uncontrolled psychological disturbances identified by current psychiatric admission
* Psychiatric consult during admission, or need for hospital appointed sitter during admission
* Non-English speakers requiring a translator
* Current corticosteroid use or corticosteroid use during the study period (including betamethasone for promoting fetal lung maturity)
* Cognitive impairment identified by medical chart review or patients requiring a legal guardian for medical decision making

Exclusion Criteria: (additional criteria for participants that will receive hydrocortisone)

* Self-reported hypersensitivity to hydrocortisone
* Inability to consent patient and administer study drug within 12 hours of a traumatic event
* Weight < 45 kilograms (kg) or >120kg
* Subjects with systemic active infections (e.g. viral, bacterial, fungal, protozoan, or helminthic)
* Subjects with uncontrolled hypertension, renal insufficiency, or decompensated congestive heart failure
* Subjects with inflammatory bowel disease
* Subjects with active or latent peptic ulcers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 133 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
PTSD assessed by the City Birth Trauma Scale | up to 6 weeks
  This is a 29 question scale that can range from 0 to 60 (a higher score indicates greater severity of symptoms of PTSD). The response scale for symptoms asks for frequency of symptoms over the last week and is scored on a scale ranging from 0 ("not at all") to 3 ("5 or more times").
  The distribution of PTSD scores will be compared between the hydrocortisone group and matched controls using appropriate statistical techniques.

SECONDARY OUTCOMES:
Mean depression scores assessed by the Edinburgh Postnatal Depression Scale19 (EPDS) | up to 6 weeks
  This is a 10 question scale and scores can range from 0 to 30. Probable postpartum depression will be defined as a score ≥ 10 and reported as Yes or No. The scores will be compared across the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna A Kountanis, MD, Principal Investigator — Assistant Professor of Anesthesiology and Assistant Professor of Obstetrics and Gynecology
Locations (1):
- Michigan Medicine - University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kountanis JA, Muzik M, Mentz G, Zhao X, Vlisides PE. Glucocorticoids after birth trauma and the associated risk of developing posttraumatic stress disorder: a non-randomized open-label pilot trial. Front Glob Womens Health. 2026 Jan 9;6:1557552. doi: 10.3389/fgwh.2025.1557552. eCollection 2025. PMID 41586417